CLINICAL TRIAL: NCT03683524
Title: Efficacy and Safety of a Simplification Strategy Based on Dolutegravir and Darunavir / Cobicistat vs Optimized Treatment in Suppressed HIV-1-infected Patients Carrying Archived Multidrug Resistance Mutations.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia (Other)
Collaborators: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Study 2D
Record Dates: First submitted 2018-07-30; First posted 2018-09-25 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: HIV-1 Infection
Keywords: Simplification strategy; Multidrug resistant; Dolutegravir; Darunavir/cobicistat; Bitherapy
MeSH Terms: interventions — dolutegravir; Cobicistat

STUDY DESIGN:
Intervention Model Description: * Experimental group: bitherapy based on DTG (50 mg QD) plus DRV/cobi (800/150 mg QD)
  * Control group: continuation of their current stable ART.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): bitherapy based on DTG (50 mg QD) plus DRV/cobi (800/150 mg QD)
  Interventions: Drug: Dolutegravir (DTG) plus Darunavir/cobicistat (DRV/cobi).
- Control group (Active Comparator): continuation of their current stable ART
  Interventions: Drug: Current ART

INTERVENTIONS:
Drug: Dolutegravir (DTG) plus Darunavir/cobicistat (DRV/cobi). — bitherapy based on DTG (50 mg QD) plus DRV/cobi (800/150 mg QD)
  Arms: Experimental group
Drug: Current ART — To continue with their current ART
  Arms: Control group

SUMMARY:
The availability of antiretroviral therapy has led to a reduction in morbidity and mortality in patients with chronic HIV infection. The treatment, however, is not free of side effects, has potential interactions with other medications, is expensive and can be complex, especially in those patients who are very experienced and with mutations that give them resistance to multiple drugs. For this reason, the development of simplification strategies that avoid unnecessary exposure to antiretroviral agents remains of great interest.

This is a simplification study, in which the investigators try to evaluate that with less medication the investigator can maintain the same virological control of the disease. This would mean a lower burden of medication for patients, facilitating its administration and reducing the number of unwanted side effects.

Specifically, the investigators intend to evaluate the treatment with Darunavir / cobicistat plus Dolutegravir as a simplification strategy, since both drugs are taken once a day, have a powerful antiviral activity, even against antiretroviral resistant viruses, and are among the best tolerated (with fewer side effects). The results reported in some observational studies suggest that two-drug therapy (bitherapy) as a simplification strategy could also be safe and effective, however, as far as the investigators know, there are no data and clinical trials that specifically evaluate darunavir / cobicistat plus dolutegravir as a strategy of simplification.

DETAILED DESCRIPTION:
The availability of antiretroviral therapy (ART) has led to a reduction in morbidity and mortality in patients with chronic HIV infection. ART, however, is not free of side effects, has potential pharmacological interactions with other drugs, is expensive and can be complex, especially in those patients with high therapeutic experience and archived antiretroviral drug resistance mutations (DRM). For this reason, the development of simplified and equally effective therapeutic strategies that save patients from exposure to antiretroviral agents remains of great interest, even in patients with DRM and limited therapeutic options.

Currently, Darunavir (DRV) in combination with either ritonavir (RTV) or cobicistat (COBI) is the most widely recommended boosted protease inhibitor. It is used in most clinical settings, including those with limited therapeutic options and highly ART-experienced patients carrying multiple DRM. In addition, DRV has good tolerance and safety profiles, a high genetic barrier and can be administered once daily in patients harboring DRM in the viral protease with little or no impact on viral sensitivity (1). As a booster, RTV has an inducing effect on glucuronidation and a broad and potent inhibitory effect on cytochrome P-450 (CYP) isozymes and drug transporters, resulting in a significant number of drug interactions. A low dose of RTV does not appear to cause substantial antiviral activity, although its theoretical contribution to the emergence of drug resistance is still unclear. By contrast, the metabolism of COBI is predominantly via CYP3A4 oxidation and, to a lesser degree, CYP2D6. COBI does not undergo glucuronidation. In addition, 99% of COBI remains unchanged, and the resulting metabolites do not seem to show any clinically relevant inhibitory activity.

Dolutegravir (DTG) is the latest available agent within the antiretroviral class of integrase strand-transfer inhibitors (INSTI). In this group, DTG is the drug with the greatest genetic barrier, derived from its greater affinity for integrase and its consequent longer dissociation time of the drug-integrase complex. The development of DTG resistance associated mutations reported in the clinical setting has been purely anecdotal, and it has not been observed in clinical trials in naïve patients. Moreover, DTG retains the ability to inhibit viral replication when integrase associated mutations have been selected by other INSTI-based treatments (i.e., raltegravir and elvitegravir/cobicistat). DTG may also favor therapeutic adherence due to its high tolerability and easy administration with once or twice daily dosages depending on the absence or presence of mutations in the integrase or prior failures with other INSTIs. Finally, DTG is eliminated mainly through metabolism by UGT1A1, and it is also a substrate of UGT1A3, UGT1A9, CYP3A4, Pgp, and BCRP. Therefore, all drugs that induce these enzymes may decrease DTG's plasma concentration and reduce its therapeutic effect. In one study, coadministration of DRV/rtv (600/100 mg twice daily) and DTG (30 mg once daily) decreased DTG Cmax, AUC and Ctrough by 11%, 22% and 38%, respectively (2). Despite these changes, it is assumed that DRV/rtv has no clinically significant effect on the pharmacokinetics of DTG and no dose adjustment is recommended.

It has been established that it is necessary to have at least two active drugs within the optimized ART to achieve and maintain virological suppression in multi-treated patients with multiple DRM. In addition, some studies have shown that recycled NRTIs or NNRTIs with residual activity are not necessary and can be withdrawn from ART optimized regimens in extensively pretreated patients with sustained virological suppression (3). In fact, limited data from some observational and clinical studies further suggest that bitherapy as simplification strategy could be also safe and effective (4). Recently, an observational study performed on a limited and heterogeneous number of highly pretreated patients who were switched to DRV/rtv plus DTG reported efficacy rates of virological suppression of up to 98% at 48 weeks (5). In addition, there are two ongoing studies (NCT02491242 and NCT02486133) that are currently evaluating bitherapy consisting of DTG and DRV. The first of these studies is an observational study with no comparator arm which is evaluating the efficacy of DTG-based bitherapy, including RPV, 3TC, or boosted DRV (both with RTV and COBI) as the second agent. The second one is a clinical study comparing the switch to DTG plus DRV/rtv vs. triple ART based on DRV/rtv in patients with limited ART experience and virological suppression. Due to the greater specificity of COBI for CYP3A4 and its lack of effect on glucuronidation in comparison to RTV, DTG plus DRV/cobi bitherapy would constitute a simplification strategy for ART consisting of two drugs with well-known efficacy, safety, tolerability, high genetic barrier, once-daily administration, and relatively less potential for pharmacological interactions than traditional optimized based regimens. As far as the investigators know, however, there are no pharmacokinetic data and clinical trials specifically evaluating DRV/cobi plus DTG as a simplification strategy.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 infected patients (≥18 years).
2. Confirmed plasma HIV-1 RNA levels < 50 copies/ml for ≥ 6 months preceding the study randomization.
3. Currently ART containing at least 3 antiretroviral drugs (protease inhibitors, non- nucleoside reverse transcriptase inhibitors, integrase inhibitors and CCR5 receptor antagonists on routine clinical practice).
4. Must have historical genotyping tests showing DRM associated with at least two antiretroviral classes according to Stanford dB.
5. Willing and able to be adherent to their cART regimen for the duration of the study (in opinion of physician).
6. If heterosexually active female; using an effective method of contraception (hormonal contraception, intra-uterine device (IUD), or anatomical sterility in self or partner*) from 14 days prior to study inclusion and at least 12 weeks after the end of the study; all female volunteers must be willing to undergo urine pregnancy tests at time points specified in the Schedule of Procedures.
7. If heterosexually active male; willing to use an effective method of contraception (anatomical sterility in self) or agree on the use of an effective method of contraception by his partner (hormonal contraception, intra-uterine device (IUD), or anatomical sterility*) from the day of the study inclusion until 12 weeks after the end of the study.
8. Signed informed consent

   * condom use nor diaphragma are considered as an additional method of contraception only and cannot be the only method of contraception used as not been considered an effective method by the Clinical Trial Facilitation Group (CTFG) guidelines.

Exclusion Criteria:

* 1. Subjects with any DRM associated to INSTI (i.e. T66I, 74M, E92Q, T97A, F121Y, E138A/K, G140A/S, Y143R/H/C, S147G, Q148H/K/R, N155H AND R263K) in historical genotyping tests. 2. Subjects with any evidence of previous virologic failure to INSTI-based regimens (with or without DRM in the integrase). 3. Subjects who have experienced previous uncontrolled interruptions of INSTI-based regimens. 4. Subjects who have archived DRM conferring a low - or higher - level of resistance to DRV/cobi (>15 points from Stanford dB score). 5. Subjects with unstable liver disease (as defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, or persistent jaundice), cirrhosis, known biliary abnormalities (apart from hyperbilirubinemia or jaundice due to Gilbert's syndrome or asymptomatic gallstones) 6. Subjects with severe hepatic impairment (class C) according to the Child-Pugh classification 7. Subjects with alanine aminotransferase (ALT) ≥ 5 times upper normal limit (ULN) or ALT ≥ 3 times ULN and bilirubin ≥ 1.5 times ULN. 8. Subjects with hepatitis C co-infection that would require therapy during the study.

  9. Subjects with hepatitis B surface antigen (HBsAg) positive. 10. Known allergy to the study drugs or their components. 11. Current or prior therapy which, in the opinion of the investigators, would make the individual unsuitable for the study or influence the results of the study. 12. Females who are pregnant or breastfeeding

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2021-08-10 (Actual); Study Completion 2021-08-10 (Actual)

PRIMARY OUTCOMES:
Plasma HIV-1 RNA < 50 copies/mL at 48 weeks | week 48
  HIV-1 RNA < 50 copies/mL using a Time to Loss of Virological Response (TLOVR).

SECONDARY OUTCOMES:
Percentage of patients developing ART-associated adverse events | Since baseline to week 48
  Percentage of patients developing ART-associated adverse events leading to treatment discontinuation.
Changes in CD4+ cell count | Since baseline to week 48
  CD4+ cell count changes
Emergence of new mutations in HIV-1 protease and integrase | Baseline and in case of virological failure, defined as ≥ 50 copies/mL in 2 consecutive determinations or a single HIV-1 RNA values > 1000 copies/mL. We can observe a virological failure throughout the study (from baseline to week 48)
  Emergence of new mutations in HIV-1 protease and integrase assessed with a genotyping test (attempted on any post Day 1 sample with HIV-1 RNA ≥ 50 copies/mL).
Plasma HIV-1 RNA < 50 copies/mL at 24 weeks | Week 24
  HIV-1 RNA< 50 copies/mL at 24 weeks by TLOVR
Plasma HIV-1 RNA < 50 copies/mL at 24 and 48 weeks | Week 24 and 48
  HIV-1 RNA < 50 copies/mL at 24 and 48 weeks using the FDA snapshot analysis (sensitivity analysis).
DTG and DRV/cobi plasma concentration | Week 4
  Description of plasmatic trough levels of DTG and DRV/cobi in the experimental group, and in those participants experiencing virological failure.
Cost associated with the antirretroviral treatment of the study | Since baseline to week 48
  ART prices
Estimated costs of clinical controls | Since baseline to week 48
  Prices of clinical controls during the study
Genotyping tests cost | At virological failure, defined as ≥ 50 copies/mL in 2 consecutive determinations or a single HIV-1 RNA values > 1000 copies/mL. We can observe a virological failure throughout the study (from baseline to week 48)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Germans Trias I Pujol, Badalona, Barcelona, Spain

REFERENCES:
- [Derived] Santos JR, Domingo P, Portilla J, Gutierrez F, Imaz A, Vilchez H, Curran A, Valcarce-Pardeiro N, Payeras A, Bernal E, Montero-Alonso M, Yzusqui M, Clotet B, Videla S, Molto J, Paredes R. A Randomized Trial of Dolutegravir Plus Darunavir/Cobicistat as a Switch Strategy in HIV-1-Infected Patients With Resistance to at Least 2 Antiretroviral Classes. Open Forum Infect Dis. 2023 Oct 31;10(11):ofad542. doi: 10.1093/ofid/ofad542. eCollection 2023 Nov. PMID 38023553